CLINICAL TRIAL: NCT03022266
Title: A Behavioral Economics-Based Telehealth Intervention to Improve Post-MI Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellth Inc. (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: W000001
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Myocardial Infarction, Acute; Myocardial Infarction
Keywords: Adherence; CleverCap® Lite BLE C035; Smartphone App; Telehealth; Digital Health; Mobile Phone App; Behavioral Economics; Aspirin; Wellth App
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants receiving the Financial Incentive and Mobile Phone App will be given an smartphone app offering pill reminders and $50/month financial incentives for three months to upload photos of medication each day for 90 days. Medication adherence will be measured via a CleverCap(R) electronic monitoring pillbox.
  Interventions: Behavioral: Financial Incentive and Mobile Phone App
- Usual Care Control Arm (No Intervention): Participants in the usual care control arm will receive the usual education about medications provided by hospital staff. Medication adherence will be measured via a CleverCap(R) electronic monitoring pillbox.

INTERVENTIONS:
Behavioral: Financial Incentive and Mobile Phone App — Subjects receiving the Financial Incentive and Mobile Phone App will each participate in a 90-day adherence promotion program. When users first log in to the app, the screen will display an incentive of $150 that participants have earned by enrolling in the program. Participants will be told that each missed medication check-in will result in a $2 deduction from the account before it is paid out. Each $50 portion (minus any penalties) of the $150 incentive will be paid out in 30-day installments by remotely crediting a previously distributed debit card. Adherence will be measured simultaneously by app photos and CleverCap(R) electronic monitoring (EM) devices filled with a 90-day supply of aspirin. Claims data will be analyzed for a 90 day period to account for any hospital admissions.
  Other Names: Smartphone App; Wellth App; Adherence; Mobile Phone App
  Arms: Intervention Arm

SUMMARY:
The proposed study is a pilot randomized clinical trial (RCT). Participants in the intervention arm will participate in a 90-day adherence promotion program based on the theory of behavioral economics and administered through the Wellth mobile phone application. Subjects will be provided a CleverCap® Lite BLE C035 smart pill bottle (electronic monitoring (EM), device) containing a 90-day supply of aspirin (90 pills) and those in the intervention arm will be offered $150 for app-based medication check-ins, which consist of uploading daily photos of pills at the time of administration through the Wellth app. Subjects will have $2 deducted from total rewards for each day that a medication check-in is missed. Subjects in the control arm will receive usual care and be monitored with the same EM device types used in the intervention arm.

DETAILED DESCRIPTION:
Medication adherence is a quantifiable parameter detailing when and how consistently doses are taken. Elements of medication adherence include: 1) the proportion of prescribed drug taken or %PDT (primary outcome); 2) the proportion of days with the correct number of doses taken; 3) the proportion of doses taken on time, in relation to a prescription-defined time interval between successive doses; 4) the distribution of inter-dose intervals; 5) the number of drug holidays; and 6) the longest interval between two doses [Vrijens et al. British journal of clinical pharmacology. 2012;73(5):691-705]. Medication adherence will be assessed in all participants using EM technology manufactured by CleverCaps®. Electronic Monitoring (EM) is more sensitive, reliable and valid than other measurement techniques such as pill counts, self-reports, or clinical judgment [Vrijens et al. Expert review of clinical pharmacology. 2014;7(5):633-644]. In this study the investigators will monitor a single drug, aspirin, in MI patients prescribed aspirin on hospital discharge.

In addition to measurement of medication adherence using an EM device, the investigators will measure adherence using the Wellth cell phone app in the intervention arm. Participants in the intervention arm will also be asked to track their medication-taking habits by uploading photos of their medications at the appropriate dosage times using the Wellth app.

Readmissions will be measured using the EMR and by interview to capture events outside the Penn system. Events will be classified according to timing (e.g. 30-day readmission) and cause (e.g. cardiac, all-cause). This study is not designed to detect a statistically significant difference in readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Over 21 years of age
* Admitted to one of the University of Pennsylvania hospitals for acute myocardial infarction (ICD-10 codes I21.xx) or unstable angina (ICD 10 codes I20.xxx)
* Prescribed once-per-day aspirin at discharge
* The patient administers his or her own medications
* Own a smartphone with a sufficient data plan or home Wi-Fi to enable app use and avoid overage charges
* Able to speak and understand English

Exclusion Criteria:

* Diagnosis of MI following non-cardiac admission
* Discharge to any facility other than the patient's home
* Cognitive impairment that limits ability to understand and complete questionnaires
* Inability to operate a mobile phone and the Wellth app
* Physician-estimated life expectancy less than 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 90 Days
  Better medication adherence at 90 days as Percentage of Doses Taken (%PDT) using CleverCap(R) electronic monitoring devices

SECONDARY OUTCOMES:
30-Day All-cause Readmissions | 30 Days
  Average rates of hospital readmissions within 30 days assessed by medical record review and patient interviews
90-Day All-cause Readmissions | 90 Days
  Average rates of hospital readmissions within 90 days assessed by medical record review and patient interviews
Medication adherence assessed using patient smartphone photos | 90 Days
  % PDT will not differ between the app and electronic monitoring measurement approaches
Self-reported self-care | 90 Days
  Self-care of coronary heart disease inventory

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Riegel, PhD, RN, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho PM, Bryson CL, Rumsfeld JS. Medication adherence: its importance in cardiovascular outcomes. Circulation. 2009 Jun 16;119(23):3028-35. doi: 10.1161/CIRCULATIONAHA.108.768986. PMID 19528344
- [Background] Zhang Y, Kaplan CM, Baik SH, Chang CC, Lave JR. Medication adherence and readmission after myocardial infarction in the Medicare population. Am J Manag Care. 2014;20(11):e498-505. PMID 25651604
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Choudhry NK, Avorn J, Glynn RJ, Antman EM, Schneeweiss S, Toscano M, Reisman L, Fernandes J, Spettell C, Lee JL, Levin R, Brennan T, Shrank WH; Post-Myocardial Infarction Free Rx Event and Economic Evaluation (MI FREEE) Trial. Full coverage for preventive medications after myocardial infarction. N Engl J Med. 2011 Dec 1;365(22):2088-97. doi: 10.1056/NEJMsa1107913. Epub 2011 Nov 14. PMID 22080794
- [Background] Jackevicius CA, Li P, Tu JV. Prevalence, predictors, and outcomes of primary nonadherence after acute myocardial infarction. Circulation. 2008 Feb 26;117(8):1028-36. doi: 10.1161/CIRCULATIONAHA.107.706820. PMID 18299512
- [Background] Ho PM, Spertus JA, Masoudi FA, Reid KJ, Peterson ED, Magid DJ, Krumholz HM, Rumsfeld JS. Impact of medication therapy discontinuation on mortality after myocardial infarction. Arch Intern Med. 2006 Sep 25;166(17):1842-7. doi: 10.1001/archinte.166.17.1842. PMID 17000940
- [Background] Choudhry NK, Avorn J, Antman EM, Schneeweiss S, Shrank WH. Should patients receive secondary prevention medications for free after a myocardial infarction? An economic analysis. Health Aff (Millwood). 2007 Jan-Feb;26(1):186-94. doi: 10.1377/hlthaff.26.1.186. PMID 17211028
- [Background] Granger BB, Bosworth HB. Medication adherence: emerging use of technology. Curr Opin Cardiol. 2011 Jul;26(4):279-87. doi: 10.1097/HCO.0b013e328347c150. PMID 21597368
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Kimmel SE, Troxel AB, Loewenstein G, Brensinger CM, Jaskowiak J, Doshi JA, Laskin M, Volpp K. Randomized trial of lottery-based incentives to improve warfarin adherence. Am Heart J. 2012 Aug;164(2):268-74. doi: 10.1016/j.ahj.2012.05.005. PMID 22877814
- [Background] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835
- [Background] Riegel B, Jaarsma T, Stromberg A. A middle-range theory of self-care of chronic illness. ANS Adv Nurs Sci. 2012 Jul-Sep;35(3):194-204. doi: 10.1097/ANS.0b013e318261b1ba. PMID 22739426
- [Background] Galloway GP, Coyle JR, Guillen JE, Flower K, Mendelson JE. A simple, novel method for assessing medication adherence: capsule photographs taken with cellular telephones. J Addict Med. 2011 Sep;5(3):170-4. doi: 10.1097/ADM.0b013e3181fcb5fd. PMID 21844832
- [Background] Patel MS, Asch DA, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults. Ann Intern Med. 2016 Oct 18;165(8):600. doi: 10.7326/L16-0280. No abstract available. PMID 27750316